CLINICAL TRIAL: NCT01561365
Title: Applicability of the Ottawa Ankle Rules to Exclude Fractures of the Ankle and Midfoot - Comparison to Orthopedic Residents Routine.
Brief Title: Applicability of the Ottawa Ankle Rules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, KANDEL, Orthopediv Surgeon, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ottawarules
Record Dates: First submitted 2012-03-18; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Ankle Fracture; Ankle Sprain
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emergency (Experimental)
  Interventions: Behavioral: Ottawa ankle rules
- Orthopedic residents (Experimental)
  Interventions: Behavioral: Ottawa ankle rules

INTERVENTIONS:
Behavioral: Ottawa ankle rules — Ottawa ankle rules implementation
  Other Names: OAR

SUMMARY:
The aim of this prospective study was to compare outcomes in patients handled by emergency physician according to OAR versus by an orthopedic resident.

92 consecutive patients with ankle injuries attending our emergency department were divided in two groups. The study group comprised 32 patients who arrived during the morning shift and were examined by an emergency physician according to OAR. Patients discharged without an x-ray were followed in the clinic or by telephone communication. The control group constituted 60 patients who were examined during the evening and night shifts by orthopedic residents unaware of this study.

DETAILED DESCRIPTION:
Objective. Ankle and midfoot injuries are common orthopedic complaints, both in general medicine and orthopedic practice. The percentage of fractures among these injuries is small, however many will undergo x-ray. Ottawa ankle rules (OAR) are clinical guidelines for determining whether to use radiography in such cases. The aim of this prospective study was to compare outcomes in patients handled by emergency physician according to OAR versus by an orthopedic resident. Also, we validated the applicability of OAR in an emergency department in our country.

Methods. 92 consecutive patients with ankle injuries attending our emergency department were divided in two groups. The study group comprised 32 patients who arrived during the morning shift and were examined by an emergency physician according to OAR. Patients discharged without an x-ray were followed in the clinic or by telephone communication. The control group constituted 60 patients who were examined during the evening and night shifts by orthopedic residents unaware of this study.

ELIGIBILITY:
Inclusion Criteria:

* ankle trauma

Exclusion Criteria:

* unwilling to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2003-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Amount of patients sent to xrays | 2 hours

SECONDARY OUTCOMES:
missed fractures | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Kandel, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel